CLINICAL TRIAL: NCT04506554
Title: A Phase II Trial of Risk Enabled Therapy After Neoadjuvant Immunochemotherapy for Bladder Cancer
Brief Title: A Study of Risk Enabled Therapy After Neoadjuvant Immunochemotherapy for Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-176; 20-1047 (Other: Fox Chase Cancer Center IRB)
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Muscle-Invasive Bladder Carcinoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMVAC + nivolumab (Experimental): This will be a single-arm, open-label, multicenter phase 2 study of neoadjuvant nivolumab with AMVAC. Approximately 70 evaluable patients will be enrolled into this study. Eligible patients will be those with diagnosis of muscle invasive urothelial carcinoma of the bladder who are cT2 or cT3 but not clinical N1 at diagnosis. Clinical stage is confirmed by transurethral resection of bladder tumor (TURBT#1).
  Interventions: Drug: AMVAC + Nivolumab

INTERVENTIONS:
Drug: AMVAC + Nivolumab — Nivolumab 240mg will be administered intravenously for 3 doses - on days 1, 15 and 29. AMVAC will be dosed intravenously every 2 weeks for 3 doses on days 1, 15 and 29 with Neulasta or equivalent. Standard AMVAC dose is as follows: methotrexate 30mg/m2, vinblastine 3mg/m2, doxorubicin 30mg/m2, and cisplatin 70mg/m2.

SUMMARY:
Neoadjuvant accelerated methotrexate/vinblastine/adriamycin/cisplatin (AMVAC) in combination with nivolumab is under evaluation for the treatment of muscle invasive bladder cancer (MIBC). Patients with pre-specified tumor mutations and complete clinical response with neoadjuvant therapy will preserve their bladders and go on active surveillance.

DETAILED DESCRIPTION:
Muscle invasive bladder cancer (MIBC) constitutes 20-25% of all cases with 5 year survival estimated at 45% regardless of treatment.1-4 Although neoadjuvant cisplatin-based chemotherapy (NAC) followed by a radical cystectomy or cystoprostatectomy with a lymph node dissection is the preferred treatment choice for MIBC in the United States, there are several drawbacks and challenges with this approach. Patients must be fit to undergo a surgical intervention. Grade 2 through 5 complications have been documented in 53% of patients undergoing cystectomy at a tertiary care center, and the surgical mortality rate is 1.5%.5, 6 Furthermore, urinary diversion commonly requires an ileal conduit and an external appliance, impacting patient's quality of life.

By incorporating neoadjuvant nivolumab with AMVAC, our goal in RETAIN-2 is to increase the number of patients who would be eligible for bladder preservation while maintaining the long-term oncologic outcomes. Nivolumab, an anti-PD1 therapy, is FDA approved for treatment of metastatic urothelial carcinoma post platinum-based chemotherapy.20 Recently, neoadjuvant pembrolizumab (anti-PD1) and atezolizumab (anti-PDL1) was tested in MIBC in the PURE-01 and ABACUS studies, and a pT0 rate of 38.6% and 29%, respectively, was achieved.21, 22 Additionally, recent work by Kim et al. presented at AACR 2019 demonstrated that AMVAC induces gene signatures in luminal tumors and may have a synergistic response with immunotherapy. Given the impressive activity of both AMVAC and nivolumab in the neoadjuvant setting, in this study the investigators hypothesize that using the combination of neoadjuvant nivolumab and AMVAC will lead to higher cT0 rate and metastasis-free survival at 2 years. At the same time by using the risk adapted strategy, a select group of patients will be able to preserve their bladders and significantly improve their quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years
* Primary urothelial or predominantly urothelial carcinoma of the bladder confirmed from pathology report. Patients with some component of variant histology mixed with predominant urothelial carcinoma will be allowed. Upper tract urothelial carcinoma patients are not allowed.
* Urothelial carcinoma of the prostatic urethra in men is allowed
* Histologic evidence of muscularis propria invasion.
* AJCC23 clinical stage T2-T3 N0M0.
* No radiographic evidence of lymph node positive disease as per RECIST 1.1 (≥15 mm short axis diameter). Lymph node positive disease is defined as clinical lymphadenopathy on staging CT or MRI greater than 1.4 cm in the short axis. If a lymph node is greater than 1.4 cm, it has to be biopsy proven negative for the patient to be eligible.
* No metastatic disease (M0).
* ECOG performance status 0, or 1.
* Left ventricular ejection fraction ≥ 50% by MUGA or ECHO within 6 months of study entry.
* Negative pregnancy test in women of child bearing potential within 24 hours of study registration. If the pregnancy test is positive, the patient must not receive protocol treatment and must not be enrolled in the study.
* Normal organ and bone marrow function (Leukocytes ≥ 3,000/mcL, Absolute neutrophil count ≥ 1,500/mcL, Platelets ≥ 100,000/mcL, Total bilirubin ≤ institutional upper limit of normal (ULN) unless patient has known Gilbert's disease, in which case an elevated bilirubin is allowed, AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN, Creatinine Clearance ≥ 50 mL/min calculated using the Cockroft-Gault formula or measured with 24 hour urine collection)

Exclusion Criteria:

* Any component of small cell histology.
* Prior systemic chemotherapy or radiation therapy for urothelial carcinoma or cytotoxic chemotherapy for another malignancy within 1 year of study entry are ineligible. Patients who received immunotherapy for non-muscle invasive bladder cancer will be excluded
* Has a known additional malignancy that has had progression or has required active treatments in the last three years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. A history of prostate cancer that was treated with surgery is acceptable, provided that the following criteria are met: Stage T2N0M0 or lower; PSA undetectable for 1 year while off androgen deprivation therapy. Patients on active surveillance for low grade prostate cancer are allowed to participate.
* Patients who have received experimental agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Methotrexate, Vinblastine, Doxorubicin or Cisplatin or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined by current oral or intravenous antibiotic therapy), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the potential for teratogenic or abortifacient effects of cytotoxic chemotherapy.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cytotoxic chemotherapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with hydronephrosis that has not been addressed with a documented assessment (i.e. normal GFR, no intervention necessary) or an intervention such as placement of a stent or nephrostomy tube.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease. Use of steroids as pre-medication for contrast allergy prior to CT scans is permitted. It is acceptable to use steroids as pre-medication for AMVAC.
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Prior treatment with CD137 agonists, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Metastasis-free survival (MFS) | 2 years
  MFS is defined as a recurrence of urothelial carcinoma that is >cN1 (more than one clinically suspicious pelvic lymph node) or surgically unresectable local recurrence (e.g., >cT4a) or M1 disease.

SECONDARY OUTCOMES:
Number of days of Overall survival | up to 5 years
  Overall Survival (OS) will be defined as the number of days from study entry to death. Individuals who are alive at last contact will be censored on the date of last contact.
Number of days of Progression free survival | up to 5 years
  Progression Free Survival (PFS) for this study will be defined as the number of days from study entry to date of first evidence of tumor progression (presence of muscle invasive disease, nodal or distant recurrence) or until death from any cause, whichever comes first. Individuals that are alive and remain free of muscle invasive disease, nodal recurrence and distant disease recurrence will be censored on the date of last clinical visit.
Number of patients erporting Toxicity of neoadjuvant nivolumab and AMVAC therapy | until 100 days after the last nivolumab/AMVAC
  Toxicity, AEs, SAEs for all patients that are associated with nivolumab or AMVAC will be collected/reported at each cycle and until 100 days after lastnivolumab/AMVAC.
  Toxicity, AEs, SAEs for the CRT arm specifically will be collected/reported as follows. Grade 1-5 toxicity at C1 (start of nivolumab/AMVAC), C2 (second cycle ofnivolumab/AMVAC), C3 (third cycle of nivolumab/AMVAC), start of chemoradiation, 1/2 completion chemoradiation, completion of chemoradiation, and up to 30 days after completion of chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Ghatalia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (4):
- United States (4):
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas